CLINICAL TRIAL: NCT02648906
Title: A Clinical Trial for an Evaluation of Choline Alfoscerate and Donepezil for Cognitive Improvements of Patients With Cerebrovascular Injury in Alzheimer Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DWB_GTM001
Record Dates: First submitted 2016-01-05; First posted 2016-01-07 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Glycerylphosphorylcholine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Choline alfoscerate (Experimental): Drug: Choline alfoscerate and Donepezil
  concomitant administration
  Interventions: Drug: Choline alfoscerate
- Placebo (Placebo Comparator): Drug: Donepezil only
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Choline alfoscerate
  Arms: Choline alfoscerate
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate efficacy and safety of Choline alfoscerate and Donepezil for cognitive improvements of patients with cerebrovascular injury in Alzheimer patients

ELIGIBILITY:
Inclusion Criteria:

1. 56~90 male and female
2. Mini-Mental State Evaluation (MMSE) between 24 and 12
3. Score ≥ 2 at the New Rating Scale for Age-related White Matter Changes (ARWMC), the rating scale of cerebral ischemic injury evaluated with MRI
4. Score 0.5, 1, 2 at CDR
5. presence of at least two of the following vascular risk factors: hypertension, diabetes, obesity, ischemic heart disease, dyslipidemia, hyperhomocysteinemia, smoking, previous cerebrovascular events and familiar history of cardio-cerebrovascular diseases.
6. donepezil 10mg from 3 months ago, dose not changed during clinical trials
7. A subject who provided written informed consent to participate in this study and cooperative with regard to compliance with study related constraints

Exclusion Criteria:

1. Subjects allergic to or sensitive to the Investigational Product or applicable ingredients
2. subject who has taken below medication 1 month before screening 1) Cholinesterase Inhibitors 2) NMDA receptor antagonists 3) blood circulation supplements 4) Acetyl-L-Carnitines 5) Nicergoline 6) Subject who has taken another medication that can affect the result of primary outcome
3. subject that can't be evaluated with ADAS-cog, MMSE, NPI, ADL, CDR, Attention Questionnaire Scale etc.
4. Asthma, COPD
5. Decompensated heart disease
6. Chronic renal failure or chronic liver disease
7. Malignant tumor
8. Subject that cant' be followed up for 12 months after Investigational drug was taken.

9 Subjects who are pregnant, lactating or who plan to be pregnant during the clinical period or females of child bearing years who do not use available contraceptive methods 10. Subject who has taken other clinical or licensed medication from another clinical trial within 30 days prior screening period 11.Other subjects who are deemed not to be appropriate for this clinical study in the discretion of investigator

Ages: 56 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2015-07; Primary Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
change of ADAS-cog score compared with Baseline | 48 weeks
  Primary outcome will be evaluated with ADAS-cog questionnaire 48 weeks after taking investigational product.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Sungnam, South Korea